CLINICAL TRIAL: NCT07167771
Title: LONGITUDINAL FOLLOW-UP STUDY TO DETERMINE THE PREDICTIVE ABILITY OF A PANEL OF BIOMARKERS IN SALIVA IN HEALTHY AND PERIODONTALLY AFFECTED PATIENTS
Acronym: FLOE_long
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 165-290725
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases
Keywords: periodontal diseases; saliva; biomarkers; prediction; periodontopathogens; interleukin 1; MMP-8
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples Samples from gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants involved in an already done cross-sectional study (code 23/481-E).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is not intervention in these patients, appart from their normal dental check-up visits.

SUMMARY:
Objective: The main aim of this longitudinal clinical study is to evaluate the predictive ability of a panel of salivary biomarkers in determining periodontal health status in 2 years follow up in a group of healthy and periodontally affected individuals.

Material and methods: In this longitudinal, observational follow-up study, patients previously enrolled in a cross-sectional study at the Periodontal Postgraduate Clinic, University Complutense of Madrid, will be re-evaluated over a 2-year period. Participants (≥18 years) will be categorized into diagnostic groups based on the 2018 classification of periodontal diseases, including periodontally healthy, gingivitis, treated periodontitis (stable/unstable), and various stages of periodontitis. The study will include follow-up visits at 1 and 2 years. At each visit, participants will undergo a comprehensive medical examination to assess age, gender, weight, height, waist circumference, blood pressure, temperature, smoking and alcohol history, systemic health, and HbA1c levels. A periodontal examination will be performed at six sites per tooth, and clinical parameters including plaque, bleeding on probing, probing depth, recession, and tooth loss will be recorded. Saliva and subgingival plaque samples will be collected for biomarker and microbiological analysis. Salivary biomarkers will be measured using multiplex immunoassays, and bacterial quantification will be performed by multiplex qPCR. Data analyses: Descriptive statistics will be used to report the clinical variables and patients will be grouped according to the pre-established diagnostic categories (periodontally healthy, gingivitis, treated periodontitis patient. In order to determine the possible statistical relationship with the medical, biochemical and microbiological variables assessed, a crude bivariate analysis will first be performed by applying a mean comparison test for quantitative variables (ANOVA) and a proportion comparison test for categorical variables (Chi-square). Subsequently, those variables identified as relevant in the crude analyses will be included as confounding and/or interaction factors in a binary logistic regression model, considering the presence of periodontitis as a response variable, in order to obtain crude and adjusted OR values, together with their corresponding 95% CIs. Based on the results obtained in the biomarker analysis, a relevant statistical analysis will be performed, taking into account all the variables collected in the study. For periodontitis cases, treatment response over time will be analyzed, with subgroup comparisons between responders and non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Participants from the cohort involved in the previous cross-sectional study (code 23/481-E).
* Adults (≥ 18-year-old)
* Being able to sign an informed consent form
* Willing to participate in this observational investigation
* Diagnosed as periodontally healthy, gingivitis, treated periodontitis patient (stable / unstable), periodontitis stages I & II, or periodontitis stages III and IV (Papapanou et al. 2023) in the previous cross-sectional study (code 23/481-E)

Exclusion Criteria:

* Patients fitting to all the above inclusion criteria will be excluded from the study if unable to attend to the study-related procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted as a 2y longitudinal, observational follow-up study, from a previous cross-sectional study (code 23/481-E). The study will be conducted at the Faculty of Dentistry University Complutense of Madrid, Spain. The research group and facilities associated with the university will serve as the primary study setting for participant recruitment, data collection, and analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Salivary biomarkers | Baseline, 1 and 2 years
  Concentrations of specific biomarkers (IL-1 and MMP-8) analyzed using multiplex commercial diagnostic tests.

SECONDARY OUTCOMES:
Age | Baseline, 1 and 2 years
  Participant's age in years.
Gender | Baseline, 1 and 2 years
  Gender
Weight | Baseline, 1 and 2 years
  Weight (kg)
Height | Baseline, 1 and 2 years
  Height (cm)
Waist circumference | Baseline, 1 and 2 years
  A measuring tape will be used, and the determination will be made above the hip bone
HbA1c | Baseline, 1 and 2 years
  Following the instructions from the manufacturer of the device (A1CNow+; Bayer) and diabetic risk questionnaire (Finn-risk)
Blood pressure | Baseline, 1 and 2 years
  The procedure will follow the recommendations in the clinical practice guidelines of the American Heart Association (AHA) {Whelton, 2018 #466}. In summary, a validated and approved blood pressure monitor (Omron M6 COMFORT IT HEM-7322U-E) will be used with the patient seated, back straight, and arms supported at heart level. After the initial measurement, there will be a 5-minute rest period before taking a second reading. The average of the two readings will be considered valid.
Temperature | Baseline, 1 and 2 years
  Participant's body temperature in degrees Celsius.
Drug, alcohol, and smoking history | Baseline, 1 and 2 years
  History of participant's drug, alcohol, and smoking habits.
Nicotine dependency | Baseline, 1 and 2 years
  Assessment of nicotine dependency using the Fagerström Test for Nicotine Dependence.
Health anamnesis | Baseline, 1 and 2 years
  Relevant systemic health information collected through a complete health history questionnaire
Presence and quantification of specific periodontal pathogens | Baseline, 1 and 2 years
  P. gingivalis, A. actinomycetemcomitans, T. forsythia detected through real time PCR analysis
Plaque index | Baseline, 1 and 2 years
  categorized as presence/absence
Bleeding on probing | Baseline, 1 and 2 years
  assessed dichotomously within 15 seconds after probing
Suppuration on probing | Baseline, 1 and 2 years
  assessed dichotomously within 15 seconds after probing
Probing depth | Baseline, 1 and 2 years
  defined as the distance in mm between the bottom of the pocket and the gingival margin
Recession | Baseline, 1 and 2 years
  defined as the distance in mm between the amelocemental boundary and the gingival margin. The sum of probing depth and recession will determine the patient's clinical attachment loss
Number of teeth lost and reason | Baseline, 1 and 2 years
  Number of teeth lost and reason

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No